CLINICAL TRIAL: NCT05773534
Title: Cross-sectional Study of Calf Muscle Perfusion Via 3D Reconstruction of Multispectral Optoacoustic Tomography in Patients With Peripheral Arterial Disease After Exercise.
Brief Title: Calf Muscle Perfusion in Patients With Intermittent Claudication by 3D-reconstruction of MSOT (MSOT_IC_3D)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ulrich Rother (Other)
Collaborators: Ph.D. Student Niklas Holzwarth, Inteligent Medical Systems, German Cancer Research Center (Unknown)
Responsible Party: Sponsor-Investigator, Ulrich Rother, PD Dr. med., University Hospital Erlangen
Organization: University Hospital Erlangen (Other)
Other Study IDs: MSOT_IC_3D
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Diagnostic Imaging; Peripheral Arterial Disease; Intermittent Claudication
Keywords: Peripheral Vascular Diseases; Peripheral Arterial Disease; Peripheral Artery Disease; PAD; Intermittent Claudication; Claudicatio intermittens; Color-Coded Duplex Sonography; CCDS; Ankle Brachial Index; ABI; Multispectral Optoacoustic Tomography; MSOT; Heel Raises; 6-minute walk test; 6MWT; Muscle Perfusion; Calf Muscle Perfusion; 3D; three-dimensional
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- healthy group: Multispectral Optoacoustic Tomography (MSOT) of the Musculus triceps surae of one leg in healthy volunteers
  Physical assessment: Pulse status / Color-Coded Duplex Sonography / Ankle-Brachial Index / 6-minute walk test (6MWT) / Continued heel raises for at least 30s
  Interventions: Diagnostic Test: MSOT
- Patients with PAD in Fontaine stage II: Multispectral Optoacoustic Tomography (MSOT) of the Musculus triceps surae of the affected leg in PAD patients in Fontaine stage II (intermittent claudication)
  Physical assessment: Pulse status / Color-Coded Duplex Sonography / Ankle-Brachial Index / 6-minute walk test (6MWT) / Continued heel raises for at least 30s
  Interventions: Diagnostic Test: MSOT

INTERVENTIONS:
Diagnostic Test: MSOT — Similar as the conventional sonography, the MSOT transducer head is placed on the skin of the examined person above the target organ. But instead of sound waves, energy is applied to the tissue via laser light, leading to constant changes of minimal expansions and contractions (thermoelastic expansion) of different tissue components or molecules. The same transducer head that releases the laser flashes can also detect the emitted ultrasound waves. In the newly configured device (Acuity Echo, iThera Medical GmbH, Munich, CE-certified), an extended spectrum of laser light can be used, enabling among others the derivation of values corresponding to hemoglobin and its oxygenation levels. As hemoglobin concentration and oxygenation status are markers for perfusion, MSOT-based imaging of these parameters could be a highly sensitive and reliable method to analyze muscle perfusion.
  Other Names: multispectral optoacoustic tomograph

SUMMARY:
The aim of the proposed study is to define independent parameters for the diagnostic assessment of the perfusion situation of the calf muscle based on 3D-reconstruction of multispectral optoacoustic tomography (MSOT) in a cross-sectional collective of patients with PAD in Fontaine stage II and a healthy control group.

DETAILED DESCRIPTION:
This is a monocentric, prospective cross-sectional study which aims to compare the 3D-reconstructed optoacoustic signals in calf muscle after a exercise in patients with PAD in Fontaine stage II and a healthy control group in order to define MSOT thresholds. MSOT data will be correlated with CCDS, ABI, maximum walking distance in 6MWT, subjectively perceived absolute walking distance in everyday life, PAD-related life quality (VASCUQOL-6) and TASC II classification in angiographic imaging (only in case angiographic imaging is available and independent from this study).

Patients with intermittent claudication will be recruited during the consulting hours of the Department of Vascular Surgery, University Hospital Erlangen. Healthy volunteers will be acquired via posters in the clinic. Following detailed information about the study and after providing written consent, relevant clinical data will be collected from the electronical patient file, if available. In addition, a thorough anamnesis interview for relevant data and CCDS would be performed. Afterwards, the 3D-reconstructed parameters will be recorded by means of longitudinal MSOT scans before and after a heel raise exercise until the occurrence of claudication pain in the calf muscle. For patients with PAD, the more affected leg is examined. In healthy volunteers, either leg is examined. ABI would be measured before and after 6MWT. All data will be adequately pseudonymized in compliance with data protection regulations before they are used for statistical analysis. The duration of the study for participants will be max. 90 minutes. The angiographic imaging will be reviewed and analyzed (if available, independently from this study and the interval between MSOT measurement being lesser than 12 months). The complete study including the validation of the data by an independent study group is expected to be finished within one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PAD in Fontaine stage II or Rutherford category 1-3 or healthy volunteers
* Adults (>18 years) who are able to give their consent

Exclusion Criteria:

* Patients with PAD in Fontaine stage I, III and IV or Rutherford category 0, 4, 5 and 6 or healthy volunteers with diabetes mellitus, chronic renal failure, claudication symptoms, abnormal ABI or non-palpable foot pulses
* People with age under 18
* Absence of written consent
* Safety concerns of the study physician (person with physical, mental or psychiatric conditions which, by the judgement of the study physician, would compromise the person's safety or the quality of the data, thereby rendering the person an ineligible candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Definition of the patient groups:
  * PAD in Fontaine stage IIa
  * PAD in Fontaine stage IIb
  Definition of the healthy control group :
  * Absence of PAD
  * Absence of diabetes mellitus
  * Absence of chronic renal insufficiency
  * No symptoms of intermittent claudication
  * ABI with values between 0.9 and 1.4 (screening examination before inclusion in the study)
  * Palpable foot pulses
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-27 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Optimal diagnostic MSOT thresholds | single time point (1 day)
  Quantitative oxygenated hemoglobin signal in 3D-reconstruction (in arbitrary units).
  [This target variable is collected non-invasively using MSOT].

SECONDARY OUTCOMES:
Difference between the corresponding 3D-reconstructed MSOT values before and after exercise | single time point (1 day)
  Difference of the values before and after exercise for hemoglobin-associated parameters derived by transcutaneous MSOT inpatients in intermittent claudication stage
Reperfusion profiles of hemoglobin-associated 3D-reconstructed MSOT parameters | single time point (1 day)
  i.e. the curves of hemoglobin-associated MSOT parameters in the first ten minutes after exercise
Correlation of acquired 3D-reconstructed MSOT parameters with the CCDS flow profiles and PSVs | single time point (1 day)
  hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT in patients with PAD in Fontaine stage II correlated with the flow profiles and PSVs of A. femoralis communis and A. poplitea determined by CCDS
Correlation of acquired 3D-reconstructed MSOT parameters with the ABI | single time point (1 day)
  hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with the ABI measurements
Correlation of acquired 3D-reconstructed MSOT parameters with relative (until the first occurrence of pain) and absolute walking distance (until the first stopping due to pain) determined during the 6MWT | single time point (1 day)
  hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with relative (until the first occurrence of pain) and absolute walking distance (until the first stopping due to pain)
Correlation of acquired 3D-reconstructed MSOT parameters with maximum walking distance in the 6MWT | single time point (1 day)
  hemoglobin-associated, 3D-reconstructed MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with the maximum walking distance in the 6MWT
Correlation of acquired 3D-reconstructed MSOT parameters with the subjectively perceived maximum walking distance in everyday life | single time point (1 day)
  hemoglobin-associated, 3D-reconstructed MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with the subjectively perceived maximum walking distance in everyday life
Correlation of acquired 3D-reconstructed MSOT parameters with the perceived PAD-specific quality of life (VASCUQOL-6 questionnaire) | single time point (1 day)
  hemoglobin-associated, 3D-reconstructed MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with the perceived PAD-specific quality of life (VASCUQOL-6 questionnaire)
Correlation of the acquired 3D-reconstructed MSOT parameters with the TASC-classification (angiography) | single time point (1 day)
  hemoglobin-associated, 3D-reconstructed MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT in patients with PAD in Fontaine stage II correlated with the TASC-classification (angiography)
Confounder analysis | single time point (1 day)
  • Correlation of all collected parameters (anamnestic, demographic, physiological) with regard to their characteristics as basic confounders for the MSOT technique

CONTACTS AND LOCATIONS:
Locations (1):
- University of Erlangen-Nuremberg (FAU), Department of Vascular Surgery, Erlangen, Bavaria, Germany

REFERENCES:
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I; ESC Scientific Document Group. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS): Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteriesEndorsed by: the European Stroke Organization (ESO)The Task Force for the Diagnosis and Treatment of Peripheral Arterial Diseases of the European Society of Cardiology (ESC) and of the European Society for Vascular Surgery (ESVS). Eur Heart J. 2018 Mar 1;39(9):763-816. doi: 10.1093/eurheartj/ehx095. No abstract available. PMID 28886620
- [Background] Lawall H, Huppert P, Espinola-Klein C, Zemmrich CS, Ruemenapf G. German guideline on the diagnosis and treatment of peripheral artery disease - a comprehensive update 2016. Vasa. 2017 Mar;46(2):79-86. doi: 10.1024/0301-1526/a000603. Epub 2017 Jan 27. PMID 28128018
- [Background] Lawall H, Diehm C, Hoffmann U, Reinecke H. [Update PAVK: Epidemiology, comorbidity and prognosis of peripheral arterial obstructive disease]. Dtsch Med Wochenschr. 2015 Dec;140(24):1798-802. doi: 10.1055/s-0041-107064. Epub 2015 Dec 1. German. PMID 26625226
- [Background] Karlas A, Masthoff M, Kallmayer M, Helfen A, Bariotakis M, Fasoula NA, Schafers M, Seidensticker M, Eckstein HH, Ntziachristos V, Wildgruber M. Multispectral optoacoustic tomography of peripheral arterial disease based on muscle hemoglobin gradients-a pilot clinical study. Ann Transl Med. 2021 Jan;9(1):36. doi: 10.21037/atm-20-3321. PMID 33553329
- [Background] Larsen ASF, Reiersen AT, Jacobsen MB, Klow NE, Nordanstig J, Morgan M, Wesche J. Validation of the Vascular quality of life questionnaire - 6 for clinical use in patients with lower limb peripheral arterial disease. Health Qual Life Outcomes. 2017 Sep 22;15(1):184. doi: 10.1186/s12955-017-0760-3. PMID 28938901
- See also: 4. Lawall, H., P. Huppert, and G. Rümenapf. Periphere arterielle Verschlusskrankheit (PAVK), Diagnostik, Therapie und Nachsorge. [S3 guideline] 2015 31.03.2021]; — https://www.awmf.org/leitlinien/detail/ll/065-003.html